CLINICAL TRIAL: NCT04692870
Title: Association Between Preoperative Shock Index and Hypotension After Spinal Anaesthesia for Non-elective Caesarean Section: A Prospective Observational Study
Brief Title: Association Between Preoperative Shock Index and Hypotension After Spinal Anaesthesia for Non- Elective Caesarean Section
Status: Completed | Type: Observational
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Shirish Silwal, Junior resident, Department of anesthesiology and critical care, BPKIHS, Nepal, B.P. Koirala Institute of Health Sciences
Other Study IDs: IRC/ 1872/ 020
Record Dates: First submitted 2020-12-26; First posted 2021-01-05 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Hypotension
Keywords: cesarean section; hypotension; spinal anesthesia; shock index; post spinal hypotension; non-elective cesarean section
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a prospective observational study done in parturient planned for non-elective caesarean section. Association between shock index (HR/SBP) and post-spinal hypotension in parturient undergoing non-elective caesarean section will be evaluated in this research.

DETAILED DESCRIPTION:
Studies have shown that early hypovolemia is insufficient to produce changes in orthostatic heart rate (HR) or systolic blood pressure (SBP). Studies have shown that Shock Index (SI) as a useful indicator for acute hypovolemia. In healthy individuals, acute blood loss less than 450 mL rarely produces abnormal HR or SBP. As, several studies have shown that relationship of baseline heart rate and systolic blood pressure in predicting post spinal hypotension, this study aims to incorporate both the parameters and attempt to develop a single effective predictor for post spinal hypotension in the form of SI.

Methodology After approval from Institutional Review committee of B.P. Koirala Institute of Health Sciences, parturient undergoing non-elective caesarian of ASA PS grade II and urgency category 2 and 3, fulfilling the inclusion criteria will be informed about the study and written consent will be obtained either in labour room or in obstetric emergency ward. During this visit patient's data that includes age, indication of caesarean section, preoperative anxiety (APAIS), gestational age, and duration of fasting, height, weight, BMI and preoperative hemoglobin concentration will be recorded.

The study will be conducted in accordance with the ethical principles of the 1964 Declaration of Helsinki and STROBE (Strengthening the Reporting of Observational studies in Epidemiology) guidelines will be followed. Before patient is shifted to the operating room (OR), ranitidine 50 mg and metoclopramide 10 mg will be administered intravenously via 18 G cannula. The patient will be shifted to operating table and standard monitors 3 lead ECG, pulse oximetry and noninvasive blood pressure will be attached. Baseline vital signs heart rate and noninvasive SBP will be recorded in operation theatre in supine position with 15° left lateral tilt before administering spinal anaesthesia. NIBP will be measured by using cuff size with width of cuff bladder covering at least 40% of arm circumference and length at least 80% and will be measured from EDAN elite V8 monitors. 3 measurements of SBP will be recorded at 1 minute interval and its mean value will be taken as baseline SBP.

Also, shock index (HR/ SBP) will be calculated before administering spinal anaesthesia. At every 1 minute interval until delivery of baby, vitals parameters HR, SBP and MAP will be measured and shock index will be calculated in each time interval. Then, the patient will be placed in sitting position. Under all aseptic precautions, 2.2 ml of 0.5% hyperbaric bupivacaine with 10 µg fentanyl will be administered in sitting position in L4- L5 or L3- L4 interspace after confirmation of free flow of CSF with 25 G Quincke's needle and drug will be injected over 20 secs. Patient will be then immediately put into supine position with a right hip wedge. A 1 L co-loading of Ringer's lactate will be administered rapidly within 10 minutes via an 18 G intravenous line after administering spinal anaesthesia. Phenylepinephrine infusion will be started at 25 microgram/min immediately after the spinal injection. The sensory level of anaesthesia will be checked using loss of cold sensation with the use of alcohol soaked cotton swabs every minute until 20 mins. Surgery will be allowed once the bilateral sensory block height at T6 is achieved. Oxygen at 40% will be administered via nasal cannula at 2-4 L/min until delivery.

Hemodynamic parameters will be recorded at following time intervals: baseline, immediately after spinal anaesthesia, every minute for the first 15 minutes after spinal injection and every 2.5 mins until end of surgery. Hypotension will be treated with phenylephrine 50 µg bolus and rapid infusion of Ringer's lactate 200 ml. If bradycardia (HR< 55/min) is associated with hypotension, IV ephedrine 6 mg will be administered. If these measures fail and bradycardia is still persistent then an IV atropine 0.5 mg will be given. Intraoperative hypertension (defined as SBP greater than 120% of the baseline reading) will be managed by stopping norepinephrine infusion. The infusion will be resumed when blood pressure returns to the upper limit of the target range i.e. 20% above baseline.After delivery of the baby, 3 IU of oxytocin will be administered IV over ≥ 30 sec followed by an infusion of 10 IU/hr (oxytocin 40 IU in 500 ml of Hartmann's solution).

The total amount of intraoperative IV fluids administered and estimated blood loss will be measured. At the conclusion of the surgery, blood loss will be estimated by cumulative measurement of the following: the volume of blood in the suction canister (and subtracting the estimated amniotic fluid from the suction chamber); visual examination of the surgical sponges.

Intraoperative use of other uterotonic agent or blood transfusion will be recorded. The attending pediatrician will assess neonatal Apgar scores at 1 and 5 minutes after delivery.

Patients will be asked to report the occurrence of intraoperative nausea Incidence of intraoperative pruritus, shivering, and dizziness will also be recorded.

The primary outcome measures will be incidence of post spinal hypotension defined as SBP < 80% of baseline reading or SBP < 100 mmHg after administering of spinal anaesthesia until delivery of baby. The secondary outcome measures will be post-delivery hypotension is defined as SBP < 80% of baseline reading or SBP < 100 mmHg observed from starting oxytocin until end of surgery.

Data collection Baseline data (gestational age, preoperative hemoglobin, preoperative anxiety, uterine incision to delivery time, hemodynamic parameters) and outcome parameters will be collected in the paper case record form and entered in windows Microsoft excel spreadsheet and will use STATA version 15.0 for analysis.

ELIGIBILITY:
Inclusion Criteria:

* All parturient at term (gestational weeks ≥ 37)
* ASA (American society of Anesthesiologist) PS (Physical status) grade II
* Category 2 and 3 of non-elective caesarean section

Exclusion Criteria:

* ASA PS Grade >2
* Pregnancy induced hypertension
* Gestational hypertension
* Known fetal abnormalities
* Contraindications to spinal anesthesia
* Multiple pregnancy
* Baseline SBP< 100 mmHg
* Intrauterine growth restriction (IUGR)
* Missing height and/ or weight data
* Stillbirth
* Height: <150 cm
* Ante-partum hemorrhage
* Cardiovascular, cerebrovascular disease, endocrine disease
* Gestational diabetes
* Failed spinal anesthesia requiring GA

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients at term undergoing emergency caesarean delivery and falling under category 2 (no immediate threat to life of pregnant women and fetus) and category 3 (requiring early delivery) according to NICE (National Institute for Clinical Excellence) guideline classification of urgency of emergency caesarean section and ASA (American society of Anaesthesiologist) PS (Physical status) grade II under spinal anesthesia will be included.
Sampling Method: Non-Probability Sample
Enrollment: 337 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Incidence of post spinal hypotension | time points between administering spinal anesthesia and until delivery of baby before starting oxytocin during surgery
  SBP < 80% of baseline reading or SBP < 100 mmHg after administering spinal anesthesia

SECONDARY OUTCOMES:
post-delivery hypotension | During surgery from starting oxytocin after delivery of baby until the end of surgery
  < 80% of baseline reading or SBP < 100 mmHg observed

CONTACTS AND LOCATIONS:
Locations (1):
- Shirish Silwal, Dharān, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yentis SM, Richards NA. Classification of urgency of caesarean section. Obstet Gynaecol Reprod Med. 2008;18(5):139-40
- [Background] Kamat LL, Jha TR, Talnikar AS, Mahevi ZM, Save MP. Effect of Ondansetron in Attenuation of Post - Spinal Hypotension in Caesarean Section : A Comparison of Two Different Doses with Placebo. J Obstet Anaesth Crit Care 2017; 7 (2):69-74
- [Background] Fitzgerald JP, Fedoruk KA, Jadin SM, Carvalho B, Halpern SH. Prevention of hypotension after spinal anaesthesia for caesarean section: a systematic review and network meta-analysis of randomised controlled trials. Anaesthesia. 2020 Jan;75(1):109-121. doi: 10.1111/anae.14841. Epub 2019 Sep 18. PMID 31531852
- [Background] Sahoo T, SenDasgupta C, Goswami A, Hazra A. Reduction in spinal-induced hypotension with ondansetron in parturients undergoing caesarean section: a double-blind randomised, placebo-controlled study. Int J Obstet Anesth. 2012 Jan;21(1):24-8. doi: 10.1016/j.ijoa.2011.08.002. Epub 2011 Nov 18. PMID 22100822
- [Background] Tang L, Tang L, Li S, Huang S, Chen L, Zhang J. Spinal anaesthesia for emergency caesarean section better using 25-gauge pencil point needle or 22-gauge cutting needle: a single centre prospective study. International Journal of research in medical sciences, 2017;10(8):12293-12300
- [Background] Somboonviboon W, Kyokong O, Charuluxananan S, Narasethakamol A. Incidence and risk factors of hypotension and bradycardia after spinal anesthesia for cesarean section. J Med Assoc Thai. 2008 Feb;91(2):181-7. PMID 18389982
- [Background] Ngan Kee WD, Khaw KS, Lau TK, Ng FF, Chui K, Ng KL. Randomised double-blinded comparison of phenylephrine vs ephedrine for maintaining blood pressure during spinal anaesthesia for non-elective Caesarean section*. Anaesthesia. 2008 Dec;63(12):1319-26. doi: 10.1111/j.1365-2044.2008.05635.x. PMID 19032300
- [Background] Sklebar I, Bujas T, Habek D. SPINAL ANAESTHESIA-INDUCED HYPOTENSION IN OBSTETRICS: PREVENTION AND THERAPY. Acta Clin Croat. 2019 Jun;58(Suppl 1):90-95. doi: 10.20471/acc.2019.58.s1.13. PMID 31741565
- [Background] Bamber JH, Dresner M. Aortocaval compression in pregnancy: the effect of changing the degree and direction of lateral tilt on maternal cardiac output. Anesth Analg. 2003 Jul;97(1):256-8, table of contents. doi: 10.1213/01.ane.0000067400.79654.30. PMID 12818977
- [Background] Campagna JA, Carter C. Clinical relevance of the Bezold-Jarisch reflex. Anesthesiology. 2003 May;98(5):1250-60. doi: 10.1097/00000542-200305000-00030. No abstract available. PMID 12717149
- [Background] McCrae AF, Wildsmith JA. Prevention and treatment of hypotension during central neural block. Br J Anaesth. 1993 Jun;70(6):672-80. doi: 10.1093/bja/70.6.672. PMID 8329261
- [Background] Bishop DG, Cairns C, Grobbelaar M, Rodseth RN. Obstetric spinal hypotension: Preoperative risk factors and the development of a preliminary risk score - the PRAM score. S Afr Med J. 2017 Nov 27;107(12):1127-1131. doi: 10.7196/SAMJ.2017.v107i12.12390. PMID 29262969
- [Background] Butwick AJ, Columb MO, Carvalho B. Preventing spinal hypotension during Caesarean delivery: what is the latest? Br J Anaesth. 2015 Feb;114(2):183-6. doi: 10.1093/bja/aeu267. Epub 2014 Jul 30. No abstract available. PMID 25080429
- [Background] Saravanan S, Kocarev M, Wilson RC, Watkins E, Columb MO, Lyons G. Equivalent dose of ephedrine and phenylephrine in the prevention of post-spinal hypotension in Caesarean section. Br J Anaesth. 2006 Jan;96(1):95-9. doi: 10.1093/bja/aei265. Epub 2005 Nov 25. PMID 16311286
- [Background] Adıyeke E. Is the Emergency Cesarean Section associated with Hypotension ? Retrospective Analysis of 80 Patients Undergoing Elective or Emergency Cesarean Section under Spinal Anesthesia. Haydarpasa Numune Medical Journal 2019;59(4):342-346
- [Background] Bishop DG. Predicting spinal hypotension during caesarean section. Southern African Journal of Anaesthesia and Analgesia. 2015 ;1181:1-4
- [Background] Frolich MA, Caton D. Baseline heart rate may predict hypotension after spinal anesthesia in prehydrated obstetrical patients. Can J Anaesth. 2002 Feb;49(2):185-9. doi: 10.1007/BF03020493. PMID 11823398
- [Background] Joshi M, Raghu K, Rajaram G, Nikhil N, Kumar S, Singh A. Baseline heart rate as a predictor of post-spinal hypotension in patients undergoing a caesarean section: An observational study. J Obstet Anaesth Crit Care. 2018;8(1):20- 23
- [Background] Kinsella SM, Norris MC. Advance prediction of hypotension at cesarean delivery under spinal anesthesia. Int J Obstet Anesth. 1996 Jan;5(1):3-7. doi: 10.1016/s0959-289x(96)80067-7. PMID 15321375
- [Background] Dahlgren G, Granath F, Wessel H, Irestedt L. Prediction of hypotension during spinal anesthesia for Cesarean section and its relation to the effect of crystalloid or colloid preload. Int J Obstet Anesth. 2007 Apr;16(2):128-34. doi: 10.1016/j.ijoa.2006.10.006. Epub 2007 Feb 5. PMID 17276668
- [Background] Nani FS, Torres ML. Correlation between the body mass index (BMI) of pregnant women and the development of hypotension after spinal anesthesia for cesarean section. Rev Bras Anestesiol. 2011 Jan-Feb;61(1):21-30. doi: 10.1016/S0034-7094(11)70003-4. PMID 21334504
- [Background] Orbach-Zinger S, Ginosar Y, Elliston J, Fadon C, Abu-Lil M, Raz A, Goshen-Gottstein Y, Eidelman LA. Influence of preoperative anxiety on hypotension after spinal anaesthesia in women undergoing Caesarean delivery. Br J Anaesth. 2012 Dec;109(6):943-9. doi: 10.1093/bja/aes313. Epub 2012 Sep 10. PMID 22964265
- [Background] Fakherpour A, Ghaem H, Fattahi Z, Zaree S. Maternal and anaesthesia-related risk factors and incidence of spinal anaesthesia-induced hypotension in elective caesarean section: A multinomial logistic regression. Indian J Anaesth. 2018 Jan;62(1):36-46. doi: 10.4103/ija.IJA_416_17. PMID 29416149
- [Background] Ohpasanon P, Chinachoti T, Sriswasdi P, Srichu S. Prospective study of hypotension after spinal anesthesia for cesarean section at Siriraj Hospital: incidence and risk factors, Part 2. J Med Assoc Thai. 2008 May;91(5):675-80. PMID 18672631
- [Background] Bishop DG, Cairns C, Grobbelaar M, Rodseth RN. Heart rate variability as a predictor of hypotension following spinal for elective caesarean section: a prospective observational study. Anaesthesia. 2017 May;72(5):603-608. doi: 10.1111/anae.13813. Epub 2017 Jan 30. PMID 28133720
- [Background] Rady MY, Nightingale P, Little RA, Edwards JD. Shock index: a re-evaluation in acute circulatory failure. Resuscitation. 1992 Jun-Jul;23(3):227-34. doi: 10.1016/0300-9572(92)90006-x. PMID 1321482
- [Background] Zarzaur BL, Croce MA, Fischer PE, Magnotti LJ, Fabian TC. New vitals after injury: shock index for the young and age x shock index for the old. J Surg Res. 2008 Jun 15;147(2):229-36. doi: 10.1016/j.jss.2008.03.025. Epub 2008 Apr 10. PMID 18498875
- [Background] Rau CS, Wu SC, Kuo SC, Pao-Jen K, Shiun-Yuan H, Chen YC, Hsieh HY, Hsieh CH, Liu HT. Prediction of Massive Transfusion in Trauma Patients with Shock Index, Modified Shock Index, and Age Shock Index. Int J Environ Res Public Health. 2016 Jul 5;13(7):683. doi: 10.3390/ijerph13070683. PMID 27399737
- [Background] Sotello D, Yang S, Nugent K. Comparison of the shock index, modified shock index, and age shock index in adult admissions to a tertiary hospital. Southwest Respir Crit Care Chronicles. 2019;7(28):18-23
- [Background] Durukan P, Ikizceli I, Akdur O, Özkan S, Sözüer EM, Avşaroǧullari L, et al. Use of the shock index to diagnose acute hypovolemia. Turkish J Med Sci. 2009;39(6):833-835
- [Background] Baraff LJ, Schriger DL. Orthostatic vital signs: variation with age, specificity, and sensitivity in detecting a 450-mL blood loss. Am J Emerg Med. 1992 Mar;10(2):99-103. doi: 10.1016/0735-6757(92)90038-y. PMID 1586423
- [Background] Birkhahn RH, Gaeta TJ, Terry D, Bove JJ, Tloczkowski J. Shock index in diagnosing early acute hypovolemia. Am J Emerg Med. 2005 May;23(3):323-6. doi: 10.1016/j.ajem.2005.02.029. PMID 15915406
- [Background] Jeon YT, Hwang JW, Kim MH, Oh AY, Park KH, Park HP, Lee Y, Do SH. Positional blood pressure change and the risk of hypotension during spinal anesthesia for cesarean delivery: an observational study. Anesth Analg. 2010 Sep;111(3):712-5. doi: 10.1213/ANE.0b013e3181e8137b. Epub 2010 Aug 4. PMID 20686012
- [Background] Yokose M, Mihara T, Sugawara Y, Goto T. The predictive ability of non-invasive haemodynamic parameters for hypotension during caesarean section: a prospective observational study. Anaesthesia. 2015 May;70(5):555-62. doi: 10.1111/anae.12992. Epub 2015 Feb 12. PMID 25676817
- [Background] Manouchehrian N, Torabi F, Shayan A, Otogara M. Investigation of effect of blood pressure and heart rate changes in different positions (lying and sitiing) on hypotension incidence rate after spinal anesthesia in patients undegoing caesarean section. International Journal of Medical Research and Health sciences; 2016; 5 (7S): 407- 412
- [Background] Pokharel K, Bhattarai B, Tripathi M, Khatiwada S, Subedi A. Nepalese patients' anxiety and concerns before surgery. J Clin Anesth. 2011 Aug;23(5):372-8. doi: 10.1016/j.jclinane.2010.12.011. PMID 21802628
- [Background] Moerman N, van Dam FS, Muller MJ, Oosting H. The Amsterdam Preoperative Anxiety and Information Scale (APAIS). Anesth Analg. 1996 Mar;82(3):445-51. doi: 10.1097/00000539-199603000-00002. PMID 8623940
- [Background] Berth H, Petrowski K, Balck F. The Amsterdam Preoperative Anxiety and Information Scale (APAIS) - the first trial of a German version. Psychosoc Med. 2007 Feb 20;4:Doc01. PMID 19742298
- [Background] Klohr S, Roth R, Hofmann T, Rossaint R, Heesen M. Definitions of hypotension after spinal anaesthesia for caesarean section: literature search and application to parturients. Acta Anaesthesiol Scand. 2010 Sep;54(8):909-21. doi: 10.1111/j.1399-6576.2010.02239.x. Epub 2010 Apr 23. PMID 20455872
- [Background] Vandenbroucke JP, von Elm E, Altman DG, Gotzsche PC, Mulrow CD, Pocock SJ, Poole C, Schlesselman JJ, Egger M; STROBE Initiative. Strengthening the Reporting of Observational Studies in Epidemiology (STROBE): explanation and elaboration. Epidemiology. 2007 Nov;18(6):805-35. doi: 10.1097/EDE.0b013e3181577511. PMID 18049195
- [Background] Heesen M, Carvalho B, Carvalho JCA, Duvekot JJ, Dyer RA, Lucas DN, McDonnell N, Orbach-Zinger S, Kinsella SM. International consensus statement on the use of uterotonic agents during caesarean section. Anaesthesia. 2019 Oct;74(10):1305-1319. doi: 10.1111/anae.14757. Epub 2019 Jul 25. PMID 31347151
- [Background] Ali Algadiem E, Aleisa AA, Alsubaie HI, Buhlaiqah NR, Algadeeb JB, Alsneini HA. Blood Loss Estimation Using Gauze Visual Analogue. Trauma Mon. 2016 May 3;21(2):e34131. doi: 10.5812/traumamon.34131. eCollection 2016 May. PMID 27626017
- [Background] Peduzzi P, Concato J, Feinstein AR, Halford TR. A18 A simulation study of the number of events per variable recommended in multivariable regression analyses. Control Clin Trials. 1993;14(5):406
- [Background] Mohta M, Aggarwal M, Sethi AK, Harisinghani P, Guleria K. Randomized double-blind comparison of ephedrine and phenylephrine for management of post-spinal hypotension in potential fetal compromise. Int J Obstet Anesth. 2016 Aug;27:32-40. doi: 10.1016/j.ijoa.2016.02.004. Epub 2016 Feb 21. PMID 27020488
- [Derived] Silwal S, Subedi A, Bhattarai B, Ghimire A. Association between preoperative shock index and hypotension after spinal anesthesia for non-elective cesarean section: a prospective cohort study. BMC Anesthesiol. 2024 Oct 23;24(1):383. doi: 10.1186/s12871-024-02766-5. PMID 39443886